CLINICAL TRIAL: NCT00768638
Title: The Renal Protective Effects of Low-dose and High-dose Atorvastatin in Patients With Glomerular Disease and Proteinuria: a Randomized Controlled Double Blinded Study
Brief Title: Study of Atorvastatin Dose Dependent Reduction of Proteinuria
Acronym: SARP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Karine Marquis, Professionnelle de recherche, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRA2580119
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin 10mg (Active Comparator)
  Interventions: Drug: Atorvastatin
- Atorvastatin 40mg (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10mg 1co id (10mg active) Placebo 40mg 1co id (40mg inactive)
  Other Names: lipitor 10mg
  Arms: Atorvastatin 10mg
Drug: Atorvastatin — Atorvastatin 40mg 1co id (40mg active) Placebo 10mg 1co id (10mg inactive)
  Other Names: lipitor 40mg
  Arms: Atorvastatin 40mg

SUMMARY:
Randomized controlled double blind study of parallel groups to evaluate the comparative effects of low-dose of atorvastatin on proteinuria in patients with stage 3 or 4 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and over
* Stage 3 or 4 chronic kidney disease (modified MDRD)
* proteinuria of > 1g/d on ACEi and/or ARB, or proteinuria of > 1g/d with intolerance or contraindication to ACEi and/or ARB
* blood pressure < 130/80 mmHg or < 140/90 mmHg in patients with five or more antihypertensive drugs
* stable renal function

Exclusion Criteria:

* rapid progression of renal failure
* immunosuppressive therapy within the past 3 months
* need a renal replacement therapy within 8 months
* definite history of chronic liver disease, or abnormal liver function
* evidence of active inflammatory muscle disease
* definite previous adverse reaction to a statin
* concurrent treatment with a contraindicated drug (fibrate, macrolide antibiotic, systemic use of imidazole or triazole antifungals, protease-inhibitors, ciclosporin)
* child bearing potential
* known to be poorly compliant with clinic visits or prescribed medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-10; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
proteinuria | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Agharazii, MD, Principal Investigator — Laval University
Locations (1):
- Hôtel-Dieu de Québec Hospital, Québec, Quebec, Canada

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702